CLINICAL TRIAL: NCT02589171
Title: Randomized Trial Evaluating Effectiveness of neoClose Abdominal Closure Device Versus Carter-Thomason Needle Passer
Brief Title: The neoClose Abdominal Closure vs Carter-Thomason Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: NeoSurgical Limited (Industry)
Responsible Party: Principal Investigator, Shinil Shah, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HSC-MS-15-0668
Record Dates: First submitted 2015-10-20; First posted 2015-10-28 (Estimated); Results first posted 2019-08-15 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Surgical Port Site Hernia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Neo Close Abdominal Closure (Experimental)
  Interventions: Device: Neo Close Abdominal Closure
- Carter Thomason Device (Active Comparator)
  Interventions: Device: Carter Thomason Device

INTERVENTIONS:
Device: Neo Close Abdominal Closure — Neo Close Abdominal Closure
  Arms: Neo Close Abdominal Closure
Device: Carter Thomason Device — Carter Thomason Device
  Arms: Carter Thomason Device

SUMMARY:
The purpose of this study is to compare the neoClose abdominal closure to the standard Carter-Thomason closure in a bariatric surgery gastric bypass population.

DETAILED DESCRIPTION:
Both the neoClose abdominal closure to the standard Carter-Thomason closure will be used to close 12 mm camera port sites and 12 mm stapler port sites upon completion of a robotic assisted laparoscopic gastric bypass. The procedure requires a 12 mm port site be placed in the midline approximately 3 cm cephalad to the umbilicus and a second 12mm port site in the right mid abdomen. Port sites will be closed as defined as the inability to palpate a fascial defect and the incision being air tight upon carbon dioxide insufflation.

ELIGIBILITY:
Inclusion Criteria:

* Morbid obesity (BMI > 35).
* Completed multimodality pre operative evaluation (Psychology, Nutrition, Support Groups).
* Approved for robotic assisted laparoscopic gastric bypass.

Exclusion Criteria:

* Previous midline laparotomy or weight loss procedure.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2016-02-12 (Actual); Primary Completion 2018-04-25 (Actual); Study Completion 2018-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shinil Shah, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Neo Close Abdominal Closure | Carter Thomason Device
Started | 35 | 35
Day 1 Follow up | 35 | 35
Week 1 Follow up | 35 | 34
Week 6 Follow up | 28 | 30
Completed | 28 | 30
Not Completed | 7 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Neo Close Abdominal Closure | Carter Thomason Device | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (12) | 45 (11) | 46 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 25 | 50
  Male | 10 | 10 | 20
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 6 | 6 | 12
  Caucasian | 26 | 25 | 51
  Hispanic | 3 | 4 | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 35 | 35 | 70

OUTCOME MEASURES:

1. Primary Outcome: Technical Effectiveness as Assessed by Number of Sutures Required to Complete Closure at the Camera Port Site
Time Frame: at the time of surgery
Population: Data were not available for 4 in the NeoClose arm and 3 in the Carter Thomason arm.
Measure: Mean (Standard Deviation); unit: number of sutures
Arm/Group | Neo Close Abdominal Closure | Carter Thomason Device
Number analyzed (Participants) | 31 | 32
number of sutures | 2 (0) | 1.84 (0.37)

2. Primary Outcome: Technical Effectiveness as Assessed by Number of Sutures Required to Complete Closure at the Stapler Port Site
Time Frame: at the time of surgery
Population: Data were not available for 5 in the NeoClose arm and 6 in the Carter Thomason arm.
Measure: Mean (Standard Deviation); unit: number of sutures
Arm/Group | Neo Close Abdominal Closure | Carter Thomason Device
Number analyzed (Participants) | 30 | 29
number of sutures | 2 (0) | 1.83 (0.38)

3. Primary Outcome: Technical Effectiveness as Assessed by the Time Required to Complete Closure at the Camera Port Site
Time Frame: at the time of surgery
Population: Data were not available for 1 in the Carter Thomason arm.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Neo Close Abdominal Closure | Carter Thomason Device
Number analyzed (Participants) | 35 | 34
seconds | 20.95 (11.73) | 33.23 (25.89)

4. Primary Outcome: Technical Effectiveness as Assessed by the Time Required to Complete Closure at the Stapler Port Site
Time Frame: at the time of surgery
Population: Data were not available for 3 in the Carter Thomason arm.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Neo Close Abdominal Closure | Carter Thomason Device
Number analyzed (Participants) | 35 | 32
seconds | 18.49 (7.79) | 28.63 (11.41)

5. Primary Outcome: Technical Effectiveness as Assessed by Depth of Needle Penetration to Complete Closure at Both the Camera Port Site and Stapler Port Site
Time Frame: at the time of surgery
Population: Data were not available for 12 participants in the NeoClose arm and 16 participants in the Carter Thomason arm. For each participant analyzed, there were needle depth data available for 1, 2, 3, or 4 stitches per participant.
Measure: Mean (Standard Deviation); unit: centimeters
Units Other Than Participants: stitch
Arm/Group | Neo Close Abdominal Closure | Carter Thomason Device
Number analyzed (Participants) | 23 | 19
Number analyzed (stitch) | 80 | 74
centimeters | 3.2 (0.93) | 4.9 (1.67)

6. Primary Outcome: Technical Effectiveness as Assessed by Number of Participants With Surgical Site Occurrences Post-Operatively
Description: Surgical site occurrences include hematoma, seroma, or infection and were assessed by physical exam.
Time Frame: immediately post op
Measure: Count of Participants; unit: Participants
Arm/Group | Neo Close Abdominal Closure | Carter Thomason Device
Number analyzed (Participants) | 35 | 35
Participants | 0 | 0

7. Primary Outcome: Technical Effectiveness as Assessed by Number of Participants With Surgical Site Occurrences Post-Operatively
Description: Surgical site occurrences include hematoma, seroma, or infection and were assessed by physical exam.
Time Frame: 1 week
Measure: Count of Participants; unit: Participants
Arm/Group | Neo Close Abdominal Closure | Carter Thomason Device
Number analyzed (Participants) | 35 | 34
Participants | 0 | 0

8. Primary Outcome: Technical Effectiveness as Assessed by Number of Participants With Surgical Site Occurrences Post-Operatively
Description: Surgical site occurrences include hematoma, seroma, or infection and were assessed by physical exam.
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Neo Close Abdominal Closure | Carter Thomason Device
Number analyzed (Participants) | 28 | 30
Participants | 0 | 0

9. Primary Outcome: Technical Effectiveness as Assessed by Number of Participants With Presence of Port Site Hernia Post-operatively
Description: Abdominal ultrasound will be used to detect port site hernia.
Time Frame: 6 weeks
Population: Data were not available for 1 in the Carter Thomason arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Neo Close Abdominal Closure | Carter Thomason Device
Number analyzed (Participants) | 28 | 29
Participants | 0 | 0

10. Secondary Outcome: Pain at the 12mm Camera Port Site as Assessed by a Visual Analog Scale
Description: Pain Score is based on a visual analog scale (VAS), with a range of 0 to 10. 0 indicates no pain and 10 indicates the most painful.
Time Frame: day 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Neo Close Abdominal Closure | Carter Thomason Device
Number analyzed (Participants) | 35 | 35
units on a scale | 0.66 (1.21) | 0.66 (1.37)

11. Secondary Outcome: Pain at the 12mm Camera Port Site as Assessed by a Visual Analog Scale
Description: as for outcome 10
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Neo Close Abdominal Closure | Carter Thomason Device
Number analyzed (Participants) | 35 | 34
units on a scale | 0.34 (0.84) | 0.74 (1.21)

12. Secondary Outcome: Pain at the 12mm Camera Port Site as Assessed by a Visual Analog Scale
Description: as for outcome 10
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Neo Close Abdominal Closure | Carter Thomason Device
Number analyzed (Participants) | 28 | 30
units on a scale | 0 (0) | 0.07 (0.37)

13. Secondary Outcome: Pain at the Stapler Port Site as Assessed by a Visual Analog Scale
Description: as for outcome 10
Time Frame: day 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Neo Close Abdominal Closure | Carter Thomason Device
Number analyzed (Participants) | 35 | 35
units on a scale | 1.03 (1.89) | 1.00 (2.25)

14. Secondary Outcome: Pain at the Stapler Port Site as Assessed by a Visual Analog Scale
Description: as for outcome 10
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Neo Close Abdominal Closure | Carter Thomason Device
Number analyzed (Participants) | 35 | 34
units on a scale | 0.40 (1.50) | 1.03 (1.60)

15. Secondary Outcome: Pain at the Stapler Port Site as Assessed by a Visual Analog Scale
Description: as for outcome 10
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Neo Close Abdominal Closure | Carter Thomason Device
Number analyzed (Participants) | 28 | 30
units on a scale | 0 (0) | 0 (0)

16. Secondary Outcome: Pain as Assessed by Number of Participants Who Took Pain Medications
Time Frame: week 1
Measure: Count of Participants; unit: Participants
Arm/Group | Neo Close Abdominal Closure | Carter Thomason Device
Number analyzed (Participants) | 35 | 34
Participants | 10 | 10

17. Secondary Outcome: Pain as Assessed by Number of Participants Who Took Pain Medications
Time Frame: week 6
Measure: Count of Participants; unit: Participants
Arm/Group | Neo Close Abdominal Closure | Carter Thomason Device
Number analyzed (Participants) | 28 | 30
Participants | 0 | 1

18. Secondary Outcome: Hospital Stay Duration
Time Frame: from the the time of hospital admission to the time of hospital discharge (about 1.29 to 2.95 days)
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Neo Close Abdominal Closure | Carter Thomason Device
Number analyzed (Participants) | 35 | 35
days | 2.12 (0.57) | 2.12 (0.83)

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Neo Close Abdominal Closure | Carter Thomason Device
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 0/35 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-02): https://cdn.clinicaltrials.gov/large-docs/71/NCT02589171/Prot_SAP_000.pdf